CLINICAL TRIAL: NCT02371525
Title: Enhancing PrEP in Community Settings (EPIC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Hektoen Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01MH095628 (NIH)
Record Dates: First submitted 2015-02-19; First posted 2015-02-25 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: adherence; prevention

ARMS (2):
- Standard of Care (No Intervention)
- Prepmate (Experimental)
  Interventions: Behavioral: Prepmate

INTERVENTIONS:
Behavioral: Prepmate — A novel multi-modal, technology-based intervention for pre-exposure prophylaxis (PrEP) adherence support .
  Arms: Prepmate

SUMMARY:
To test the effectiveness of Prepmate, a novel multi-modal, technology-based intervention for pre-exposure prophylaxis (PrEP) adherence support among young men who have sex with men (MSM).

ELIGIBILITY:
Inclusion Criteria:

* HIV-uninfected as determined by a negative/non-reactive laboratory test within 7 days of Enrollment (as defined in the study-specific procedures (SSP) Manual).
* Interested in initiating PrEP
* Eligible to initiate PrEP

  * Creatinine clearance > 60 ml/min as estimated by the Cockcroft-Gault equation within 6 weeks of enrollment
  * Hepatitis B surface antigen (HBsAg) negative within 6 weeks Enrollment
  * No other medical contraindications to PrEP
* Age 18 years - 29 years
* Willing and able to provide written informed consent
* Report having had anal sex with a man in the previous 6 months
* Meet any of the following risk criteria for the prior 6 months:

  * Any condomless anal sex
  * Three or more anal sex partners
  * Self-reported new STI
  * Known HIV-infected sex partner
* Have regular access to a computer and/or a smart phone to access the internet and/or apps
* Have the ability to send and receive text messages
* Able to read and speak in English

Exclusion Criteria:

* PrEP use within the past year (PrEP naïve participants will be prioritized).
* Any reactive or positive HIV test at Screening, even if subsequent testing indicates that the person is HIV-uninfected
* Prior or current participation in the active arm of an HIV vaccine trial
* At Enrollment, has any other condition that, based on the opinion of the investigator or designee, would preclude provision of informed consent, make participation in the project unsafe, complicate interpretation of outcome data, or otherwise interfere with achieving the project objectives.
* Signs or symptoms of acute HIV infection (as described in the SSP Manual)
* History of pathological bone fracture not related to trauma.

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
PrEP adherence among young MSM over time based on dried blood spot (DBS) | DBS measured through week 36
  PrEP adherence during follow-up based on dried blood spot (DBS) concentrations.

SECONDARY OUTCOMES:
Change in PrEP knowledge assessed via computer-assisted self-interview (CASI) | baseline and week 36
  Change in PrEP knowledge assessed via computer-assisted self-interview (CASI) at baseline and week 36 (or early termination)
Change in risk behaviors administered via CASI | baseline through week 36
  Change in self-reported sexual risk behavior administered via CASI
Change in risk perception administered by CASI | baseline through week 36
  Changes in risk perception during the study administered by CASI
Acceptability of Prepmate as measured by an acceptability index collected via CASI | Month 9 (or early termination)
  Acceptability of Prepmate as measured by an acceptability index collected via CASI at 9 months (or early termination).
Perceptions of Prepmate provided via individual exit interviews | Month 10
  Qualitative feedback provided via individual exit interviews with a subset of participants one month after Prepmate termination. Interviews will be open-ended and will cover topics such as usability, acceptability, user-experience and effectiveness of the Prepmate intervention.
Patterns of use of Prepmate texting service over time as measured by responses to text messages. | through week 36
  Use patterns of Prepmate texting service over time as measured by responses to text messages.
The incidence of sexually-transmitted infection (STI) among all participants. | through week 36
  Incidence of a combination endpoint of gonorrhea, chlamydia, and/or syphilis.
The number of participants who acquire HIV | week 36
  The number of HIV infections (2) The drug resistance profiles of breakthrough infections

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Stroger Hospital and the CORE Center, Chicago, Illinois, United States

REFERENCES:
- [Derived] Liu AY, Vittinghoff E, von Felten P, Rivet Amico K, Anderson PL, Lester R, Andrew E, Estes I, Serrano P, Brothers J, Buchbinder S, Hosek S, Fuchs JD. Randomized Controlled Trial of a Mobile Health Intervention to Promote Retention and Adherence to Preexposure Prophylaxis Among Young People at Risk for Human Immunodeficiency Virus: The EPIC Study. Clin Infect Dis. 2019 May 30;68(12):2010-2017. doi: 10.1093/cid/ciy810. PMID 30239620